CLINICAL TRIAL: NCT00780091
Title: Evaluation of Efficacy and Cost of Two Monitoring Strategies for Public Clinical Research - OPTIMON: Optimisation of Monitoring for Clinical Research Studies
Brief Title: Optimisation of Monitoring for Clinical Research Studies
Acronym: OPTIMON
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Jean-Pierre LEROY / Clinical Research and Innovation Director, University hospital, Bordeaux
Other Study IDs: CHUBX 2005/04
Record Dates: First submitted 2008-05-21; First posted 2008-10-27 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: optimization; risk scale; non inferiority; cluster randomization; monitoring strategies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: classical monitoring strategy
  Interventions: Other: classical monitoring strategy
- 2: optimized monitoring strategy
  Interventions: Other: optimized monitoring strategy

INTERVENTIONS:
Other: classical monitoring strategy — intensive on-site monitoring, consistently with the pharmaceutical industry practices
  Groups: 1
Other: optimized monitoring strategy — optimized on-site monitoring, depending on patient's risk
  Groups: 2

SUMMARY:
OPTIMON will compare the efficacy and the cost of two monitoring strategies: one based on the classic standards of quality assurance, and the other one being a priori "optimized" on the main scientific and regulatory principles.

DETAILED DESCRIPTION:
There is no validated standard of monitoring strategy for clinical research studies. Optimon will compare two monitoring strategies - a classical strategy based on the practices of the pharmaceutical industry, and an optimized strategy based on patient's risk level - on their ability to produce exact data, focusing on the main quality criteria: regulatory requirements and scientific validity of results. Optimon is a non inferiority randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Research Studies: risk level A, B, or C in the Optimon risk-assessment scale, with or without a sponsor and the advice of an ethical committee, starting in 2008 and ending before the end of 2010, with a foreseen accrual of 20 patients or more, multicentric with at least 4 clinical sites, with a paper or electronic CRF, with the participating agreement of the coordinating investigator and the sponsor.
* Clinical sites: Sites with a foreseen accrual of 5 patients at least, with the participating agreement of the principal investigator.
* Clinical Research Units: with the label of an institution, with at least 2 years of experience in multicentric studies, with SOPs finalized before 2008, willing to participate in Optimon.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All type of patients enrolled in the eligible studies
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients' file without severe error. | at end of follow-up

SECONDARY OUTCOMES:
Compounds of the main outcome, other errors, delay to get the results, costs | at end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, MD, PhD, Study Director — University Hospital, Bordeaux
Locations (1):
- Unité de Soutien Méthodologique à la Recherche Clinique et Epidémiologique du CHU de Bordeaux, Bordeaux, France

REFERENCES:
- [Background] Lienard JL, Quinaux E, Fabre-Guillevin E, Piedbois P, Jouhaud A, Decoster G, Buyse M; European Association for Research in Oncology. Impact of on-site initiation visits on patient recruitment and data quality in a randomized trial of adjuvant chemotherapy for breast cancer. Clin Trials. 2006;3(5):486-92. doi: 10.1177/1740774506070807. PMID 17060222